CLINICAL TRIAL: NCT04692597
Title: Low Level Laser Therapy (LLLT) for the Treatment of Hand Osteoarthritis.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: David Moss (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Moss, Principal Investigator, Mike O'Callaghan Military Hospital
Organization: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWH20210010H
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Low Level Laser Therapy; Osteoarthritis; Family Medicine; Pain Management; Integrative Medicine
MeSH Terms: conditions — Osteoarthritis; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (LLLT) (Experimental): Group 1: Low level laser therapy (LLLT) using Phoenix Thera-lase device (74 Watts, 1275 nm wavelength) for 6 minutes affected per hand.
  The protocol for each group will involve one minute of LLLT over each of the following treatment zones: dorsal fingers and thumb, dorsal metacarpals, dorsal wrist, palmar fingers and thumb, palmar metacarpals, palmar wrist for a total of 6 minutes affected on each hand. The LLLT device will be held approximately 12 inches from the skin surface.
  Interventions: Device: Phoenix Thera-Lase System
- Group 2 (LLLT Sham) (Sham Comparator): Group 2: Sham LLLT using the Phoenix Thera-lase device with the guide light on but without emitting laser photons for 6 minutes affected per hand.
  The protocol for each group will involve one minute of sham LLLT over each of the following treatment zones: dorsal fingers and thumb, dorsal metacarpals, dorsal wrist, palmar fingers and thumb, palmar metacarpals, palmar wrist for a total of 6 minutes affected on each hand. The LLLT device will be held approximately 12 inches from the skin surface.
  Interventions: Device: SHAM Phoenix Thera-Lase System

INTERVENTIONS:
Device: Phoenix Thera-Lase System — Low level laser therapy (LLLT) using Phoenix Thera-lase device (74 Watts, 1275 nm wavelength) for 6 minutes per affected hand.
  Arms: Group 1 (LLLT)
Device: SHAM Phoenix Thera-Lase System — Sham LLLT using the Phoenix Thera-lase device with the guide light on but without emitting laser photons for 6 minutes per affected hand.
  Arms: Group 2 (LLLT Sham)

SUMMARY:
This study is a randomized, control trial of Active Duty and DoD Beneficiaries, age 18 years or older, with complaints of hand osteoarthritis. Subjects will be randomized into one of two groups receiving either LLLT or sham LLLT. Subjects will receive LLLT or sham LLLT weekly over a period of six weeks. At each visit, patients will rate their pain using the Defense and Veterans Pain Rating Scale (DVPRS) and assess their functionality using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. Subjects will have a follow up visit six weeks after the treatment protocol for a final assessment of pain and function. The Phoenix Thera-Lase laser is a Class II, 510k cleared device (#K151521) and is legally marketed in the US. Investigators are using in accordance with its approved labeling and no changes to the approved labeling are being sought.

DETAILED DESCRIPTION:
This study is a randomized, control trial of Active Duty and DoD Beneficiaries, age 18 years or older, with complaints of hand osteoarthritis. Subjects will be randomized into one of two groups receiving either LLLT or sham LLLT. Subjects will receive LLLT or sham LLLT weekly over a period of six weeks. At each visit, patients will rate their pain using the Defense and Veterans Pain Rating Scale (DVPRS) and assess their functionality using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire. Subjects will have a follow up visit six weeks after the treatment protocol for a final assessment of pain and function. The Phoenix Thera-Lase laser is a Class II, 510k cleared device (#K151521) and is legally marketed in the US. Investigators are using in accordance with its approved labeling and no changes to the approved labeling are being sought.

The Phoenix Thera-Lase System is intended to emit energy in the infrared spectrum to provide topical heating for the purpose of elevating tissue temperature for temporary relief of minor muscle and joint pain, muscle spasm, pain and stiffness associated with minor arthritis, promoting relaxation of muscle tissue and to temporarily increase local blood circulation. It is specifically designed as a high-power laser with an output power of 35 Watts and an output wavelength of1064 nm. The study will be utilizing an output power of 74 Watts and an output wavelength of 1275 nm.

ELIGIBILITY:
**Patients must be able to get care at Nellis Air Force Base (a military installation) in order to participate in this study**

Inclusion Criteria:

* Male and Female Active Duty and DoD Beneficiaries aged 18 years or older
* Hand pain, aching, or stiffness

And at least 3 of the 4 following features:

* Hard tissue enlargement of 2 or more of 10 selected joints
* Hard tissue enlargement of 2 or more distal interphalangeal (DIP) joints
* Fewer than 3 swollen metacarpophalangeal (MCP) joints
* Deformity of at least 1 of 10 selected joints

(The 10 selected joints are the first carpometacarpal (CMC), second and third proximal interphalangeal (PIP), second and third DIP joints of both hands.)

Exclusion Criteria:

* Known diagnosis of another type of arthritis: rheumatoid, psoriatic, crystalline, inflammatory bowel associated arthritis
* History of treatment with LLLT in the past 12 weeks Surgery within the past 6 weeks
* Hand fracture within the past 6 weeks
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Defense and Veterans Pain Rating Scale | visit 1 (Day 1) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 2 (Week 1) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 3 (Week 3) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 4 (Week 4) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 5 (Week 5) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 6 (Week 6) pre-treatment and immediately post-treatment *change same visit
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Defense and Veterans Pain Rating Scale | visit 7 (Week 12)
  The DVPRS consists of an 11-point numerical rating scale with 0 indicating no pain and 10 indicating severe pain. It has been confirmed for reliability and validity in measuring both acute and chronic pain, and is currently the standard for pain measurement throughout DoD and VA health systems. The DVPRS has demonstrated linear scale qualities allowing parametric methods to be used
Disabilities of the Arm, Shoulder, and Hand | visit 1 (day1) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 2 (week 2) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 3 (week 3) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 4 (week 4) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 5 (week 5) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 6 (week 6) pre-treatment and immediately post-treatment *change same visit
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Disabilities of the Arm, Shoulder, and Hand | visit 7 (week 12)
  The DASH is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point likert scale with 1 being no difficulty and 5 bring unable to perform the activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Mike O'Callaghan Military Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan on sharing data.

REFERENCES:
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Zhang W, Doherty M, Leeb BF, Alekseeva L, Arden NK, Bijlsma JW, Dincer F, Dziedzic K, Hauselmann HJ, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Maheu E, Martin-Mola E, Pavelka K, Punzi L, Reiter S, Sautner J, Smolen J, Verbruggen G, Zimmermann-Gorska I. EULAR evidence based recommendations for the management of hand osteoarthritis: report of a Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics (ESCISIT). Ann Rheum Dis. 2007 Mar;66(3):377-88. doi: 10.1136/ard.2006.062091. Epub 2006 Oct 17. PMID 17046965
- [Background] Brosseau L, Wells G, Marchand S, Gaboury I, Stokes B, Morin M, Casimiro L, Yonge K, Tugwell P. Randomized controlled trial on low level laser therapy (LLLT) in the treatment of osteoarthritis (OA) of the hand. Lasers Surg Med. 2005 Mar;36(3):210-9. doi: 10.1002/lsm.20137. PMID 15704096
- [Background] Baltzer AW, Ostapczuk MS, Stosch D. Positive effects of low level laser therapy (LLLT) on Bouchard's and Heberden's osteoarthritis. Lasers Surg Med. 2016 Jul;48(5):498-504. doi: 10.1002/lsm.22480. Epub 2016 Feb 2. PMID 26833862
- [Background] Hegedus B, Viharos L, Gervain M, Galfi M. The effect of low-level laser in knee osteoarthritis: a double-blind, randomized, placebo-controlled trial. Photomed Laser Surg. 2009 Aug;27(4):577-84. doi: 10.1089/pho.2008.2297. PMID 19530911
- [Background] Rayegani SM, Raeissadat SA, Heidari S, Moradi-Joo M. Safety and Effectiveness of Low-Level Laser Therapy in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. J Lasers Med Sci. 2017 Summer;8(Suppl 1):S12-S19. doi: 10.15171/jlms.2017.s3. Epub 2017 Aug 29. PMID 29071029
- [Background] Huang Z, Chen J, Ma J, Shen B, Pei F, Kraus VB. Effectiveness of low-level laser therapy in patients with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Sep;23(9):1437-1444. doi: 10.1016/j.joca.2015.04.005. Epub 2015 Apr 23. PMID 25914044
- [Background] Brosseau L, Welch V, Wells G, Tugwell P, de Bie R, Gam A, Harman K, Shea B, Morin M. Low level laser therapy for osteoarthritis and rheumatoid arthritis: a metaanalysis. J Rheumatol. 2000 Aug;27(8):1961-9. PMID 10955339
- [Background] Polomano RC, Galloway KT, Kent ML, Brandon-Edwards H, Kwon KN, Morales C, Buckenmaier C' 3rd. Psychometric Testing of the Defense and Veterans Pain Rating Scale (DVPRS): A New Pain Scale for Military Population. Pain Med. 2016 Aug;17(8):1505-19. doi: 10.1093/pm/pnw105. Epub 2016 Jun 6. PMID 27272528
- [Background] Nassif TH, Hull A, Holliday SB, Sullivan P, Sandbrink F. Concurrent Validity of the Defense and Veterans Pain Rating Scale in VA Outpatients. Pain Med. 2015 Nov;16(11):2152-61. doi: 10.1111/pme.12866. Epub 2015 Aug 8. PMID 26257151
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Dixon D, Johnston M, McQueen M, Court-Brown C. The Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) can measure the impairment, activity limitations and participation restriction constructs from the International Classification of Functioning, Disability and Health (ICF). BMC Musculoskelet Disord. 2008 Aug 20;9:114. doi: 10.1186/1471-2474-9-114. PMID 18715495
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Sloman R, Wruble AW, Rosen G, Rom M. Determination of clinically meaningful levels of pain reduction in patients experiencing acute postoperative pain. Pain Manag Nurs. 2006 Dec;7(4):153-8. doi: 10.1016/j.pmn.2006.09.001. PMID 17145489
- [Background] MacDermid JC, Wessel J, Humphrey R, Ross D, Roth JH. Validity of self-report measures of pain and disability for persons who have undergone arthroplasty for osteoarthritis of the carpometacarpal joint of the hand. Osteoarthritis Cartilage. 2007 May;15(5):524-30. doi: 10.1016/j.joca.2006.10.018. Epub 2006 Dec 11. PMID 17161960
- [Background] Vermeulen GM, Brink SM, Sluiter J, Elias SG, Hovius SE, Moojen TM. Ligament reconstruction arthroplasty for primary thumb carpometacarpal osteoarthritis (weilby technique): prospective cohort study. J Hand Surg Am. 2009 Oct;34(8):1393-401. doi: 10.1016/j.jhsa.2009.06.019. Epub 2009 Sep 6. PMID 19733982
- [Background] Holm, S. 1979. A simple sequential rejective multiple test procedure. Scand. J. Statistics, 6: 65-70.
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. 2016